CLINICAL TRIAL: NCT02674503
Title: Impact of a Hospital Mobility Program on Function After Discharge
Brief Title: Impact of a Mobility Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E1995-R
Record Dates: First submitted 2016-01-08; First posted 2016-02-04 (Estimated); Results first posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-03

CONDITIONS: Hospitalization
Keywords: Walking; Hospitalization; Randomized controlled trial
MeSH Terms: interventions — Walking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intensive (Experimental): MP patients will participate in a program of progressive walking and transfer training up to three times a day, seven days a week throughout the hospital stay.
  Interventions: Behavioral: Walking
- Friendly visit (Placebo Comparator): UC patients will receive three times a day "friendly visits", seven days a week by members of the research team to control for the daily attention that MP patients receive.
  Interventions: Behavioral: Friendly visit

INTERVENTIONS:
Behavioral: Walking — MP patients will participate in a program of progressive walking and transfer training up to three times a day, seven days a week throughout the hospital stay. MP patients will begin with assisted sitting, then standing, progressing to weight shifting and stepping in place, and then to walking as tolerated. The level of mobility recommended to the MP patient by the Walker will be dependent on the individual patient and will incorporate the activities patients were deemed able to do independent of cueing or assistance during each walking session.
  Arms: Intensive
Behavioral: Friendly visit — UC patients will receive three times a day "friendly visits", seven days a week by members of the research team to control for the daily attention that MP patients receive.
  Arms: Friendly visit

SUMMARY:
After hospitalization, many older adults experience more difficulty getting around in the community and performing one or more of their basic activities of daily living (ADLs) like bathing or dressing. The goals of this study are to test the effectiveness of a mobility intervention, compared to usual care, on change in mobility after hospitalization, to determine the impact on one-year outcomes such as nursing home placement and to identify which Veterans benefit the most from the intervention. Ultimately, the goal is to improve recovery after hospitalization and reduce disability in hospitalized Veterans.

DETAILED DESCRIPTION:
For this high impact study the investigators propose to use a stepped wedge cluster randomization design on five VA hospital wards to compare a mobility program (MP) to usual care (UC) among a cohort of Veterans age 50 years. The investigators will examine pre to post-hospital mobility and adverse outcomes including functional decline, nursing home admission, emergency department (ED) visits, hospitalization and death in the MP and UC groups in the year after hospital discharge. The primary outcome of mobility will be measured by the University of Alabama at Birmingham (UAB) Life-Space Assessment (LSA).10-13 Secondary measures of mobility will include self-reported ability to walk mile and drive a car, as described by Gill, et al.14 The investigators will identify patient specific characteristics that modify the effect of the mobility intervention on post-hospital mobility and adverse outcomes to determine which hospitalized patients are most likely to benefit from this intervention.

Note, Secondary outcome measures were curtailed as the original PI, Dr. Brown, retired.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 years admitted to one of the five hospital wards of the Birmingham VA Medical Center (VAMC) for any medical illness, e.g.:

  * Pneumonia
  * Heart failure
  * Chronic obstructive pulmonary disease (COPD) exacerbation
  * Or other medical (versus surgical) indication for hospitalization
* Patients will be recruited within 48 hours of hospitalization, followed throughout their hospitalization and for one year after hospital discharge.

Exclusion Criteria:

* Patients admitted for brief observation will be excluded, e.g.:

  * 23-hour observation for possible myocardial infarction
  * Additional exclusion criteria will include:
  * Inability to walk across a small room 2 weeks prior to admission
  * Inability to walk safely with assistance, based on a strength and balance screen (see Training of Walkers, below for details)
  * Having a pulmonary embolus, unstable angina or other medical diagnosis deemed by the primary physician to be a contraindication to walking
  * Being on hospice or comfort care
  * Being in a semi-private room with another currently enrolled participant
  * Non-English speaking, blind, or deaf

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2016-12-12 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia J Brown, MD MSPH, Principal Investigator — Birmingham VA Medical Center, Birmingham, AL
Locations (2):
- United States (2):
  - Birmingham VA Medical Center, Birmingham, AL, Birmingham, Alabama
  - UAB Hospital, Birmingham, Alabama

IPD SHARING:
Plan to Share IPD: Yes
No detailed plans at this time.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment were 12/12/2016 through 10/19/2019. Participant recruited from the inpatient hospital setting.
Pre-assignment Details: No significant events in the study that occurred after participant enrollment.
Period: Overall Study
Arm/Group | Intensive | Friendly Visit
Started | 62 | 70
Completed | 60 | 68
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Population: 2 participants in each group did not get randomized, n=4 without baseline data
Groups:
- Total: Total of all reporting groups
Arm/Group | Intensive | Friendly Visit | Total
Number analyzed (Participants) | 60 | 68 | 128
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.2 (8.5) | 66.2 (9.5) | 66.2 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 5 | 15
  Male | 50 | 63 | 113
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 56 | 66 | 122
  Unknown or Not Reported | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 25 | 26 | 51
  White | 30 | 38 | 68
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 60 | 68 | 128
Life Space Total Score, mean (SD) [Mean (Standard Deviation); unit: units on a scale] — The range in scores is 0-100 with higher scores representing better life space mobility. Population: Missing data on n=1 for this measure; not able to calculate score due to missing data
  units on a scale
    number analyzed (Participants) | 60 | 67 | 127
    (all) | 60.1 (28.3) | 66.5 (23.2) | 63.5 (25.8)
Activities of Daily Living Score, mean (SD) [Mean (Standard Deviation); unit: units on a scale] — Scores range from 0-12, with lower scores representing better independence in activities of daily living. Population: Missing data on n=18 for this measure; not able to calculate score due to missing data
  units on a scale
    number analyzed (Participants) | 52 | 58 | 110
    (all) | 7.5 (1.3) | 7.6 (1.8) | 7.5 (1.6)
Instrumental Activities of Daily Living Score, mean (SD) [Mean (Standard Deviation); unit: units on a scale] — A summary score ranges from 3 to 24, with higher scores indicating higher levels of independence with the tasks. Score options were trichotomous (1 = unable, 2 = needs assistance, 3 = independent).
  units on a scale | 14.7 (2.4) | 14.9 (2.2) | 14.8 (2.3)

OUTCOME MEASURES:

1. Primary Outcome: Life-Space Assessment Score
Description: The UAB Study of Aging Life-Space Assessment (LSA) is a validated tool that measures mobility and function based on the distance which a person reports moving during the four weeks preceding the assessment. The range in scores is 0-100 with higher scores representing better life space mobility.
Time Frame: One year
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intensive | Friendly Visit
Number analyzed (Participants) | 40 | 41
score on a scale | 57.8 (26.7) | 59.6 (23.3)
Statistical Analysis 1: Comparison: Intensive vs Friendly Visit; Test type: Superiority; p = 0.02, Regression, Linear — Linear fixed effect models adjusted for time in months

2. Secondary Outcome: Presence of Adverse Outcomes: Rehospitalization
Description: To determine the impact of participation in the mobility program on adverse outcomes, the investigators will measure the frequency of rehospitalization in the MP versus UC groups.
Time Frame: One Year
Reporting Status: Not Posted

3. Secondary Outcome: Presence of Adverse Outcomes: Nursing Home Placement
Description: To determine the impact of participation in the mobility program on adverse outcomes, the investigators will measure the frequency of nursing home placement in the MP versus UC groups.
Time Frame: One year
Reporting Status: Not Posted

4. Secondary Outcome: Presence of Adverse Outcomes: Death
Description: To determine the impact of participation in the mobility program on adverse outcomes, the investigators will measure the frequency of death in the MP versus UC groups.
Time Frame: One year
Reporting Status: Not Posted

5. Secondary Outcome: Activities of Daily Living (ADLs)
Description: Participants will be asked to complete the Katz ADL. Specifically, patients will be asked to rate their current level of independence with six activities of daily living (feeding, bathing, dressing, toileting, transferring, and walking across a small room). Scores range from 0-12, with lower scores representing better independence in activities of daily living.
Time Frame: One Year
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intensive | Friendly Visit
Number analyzed (Participants) | 40 | 41
score on a scale | 7.34 (0.97) | 7.37 (0.76)
Statistical Analysis 1: Comparison: Intensive vs Friendly Visit; Test type: Superiority; p = 0.13, Regression, Linear; Linear effects model adjusted for time (in months)

6. Secondary Outcome: Presence of Adverse Outcomes (ED Visits, Rehospitalization, Nursing Home Placement, Death)
Description: To determine the impact of participation in the mobility program on adverse outcomes, the investigators will measure the frequency of ED visits, hospitalizations as well as death and nursing home admissions including both short and long term placement in the MP versus UC groups.
Time Frame: One year
Reporting Status: Not Posted

7. Secondary Outcome: Instrumental Activities of Daily Living (IADLs)
Description: Level of independence with Instrumental Activities of Daily Living (IADLs) will be assessed at the same time points as the basic ADLs using the Lawton Index. The IADL index evaluates 8 domains of function including shopping, food preparation, housekeeping, laundry, transportation, handling finances, ability to take own medications and use of the telephone. A summary score ranges from 3 to 24, with higher scores indicating higher levels of independence with the tasks. Score options were trichotomous (1 = unable, 2 = needs assistance, 3 = independent).
Time Frame: One year
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intensive | Friendly Visit
Number analyzed (Participants) | 40 | 41
score on a scale | 14.0 (3.32) | 14.8 (1.96)
Statistical Analysis 1: Comparison: Intensive vs Friendly Visit; Test type: Superiority; p = 0.02, Regression, Linear; Linear mixed effects models adjusted for time (in months)

8. Secondary Outcome: Mini Cognitive Assessment (Mini-Cog)
Description: The Mini-Cog is a brief cognitive screening measure that includes a three-item memory recall and a clock drawing test. The test is scored using a simple algorithm whereby patients who are unable to recall any of the three items are considered demented; those who can recall all three items are deemed not demented; and those with intermediate word recall ability (1 or 2 items) are classified based on the clock drawing test. For persons with intermediate recall ability, if the clock drawing is abnormal, the patient is considered demented and if the clock drawing is normal the patient is not considered demented.
Time Frame: Baseline only
Reporting Status: Not Posted

9. Secondary Outcome: Confusion Assessment Method
Description: The Confusion Assessment Method (CAM) allows rapid assessment of the presence of delirium. Four clinical features, including 1) Acute onset and fluctuating course; 2) Inattention; 3) Disorganized thinking; and 4) Altered level of consciousness, are assessed. The presence of features 1 and 2 and either 3 or 4 indicates the patient has delirium. The positive and negative predictive values for the CAM are approximately 90%.
Time Frame: Baseline only
Reporting Status: Not Posted

10. Secondary Outcome: Patient Health Questionnaire (PHQ) -2
Description: Patients will be asked at each interview the Patient Health Questionnaire (PHQ) - 2, specifically 1) Have you often been bothered by feeling down, depressed, or hopeless?; and 2) Have you often been bothered by little interest or pleasure in doing things? The PHQ-2 has been found to have a sensitivity and specificity of 83% and 92% respectively and is an excellent brief screening tool for depression.
Time Frame: One year
Reporting Status: Not Posted

11. Secondary Outcome: EuroQOL Five Dimensions Questionnaire (EQ-5D)
Description: Patients will be asked to complete the EQ-5D once during the hospital stay, then at months 1, 3, 6, 9, and 12. The EQ-5D-3L is a well-validated measure of quality of life which enables the calculation of a single index value ranging from 0, worst imaginable health to 1, perfect health.
Time Frame: One year
Reporting Status: Not Posted

12. Secondary Outcome: Lubben Social Network Scale (LSNS-Revised)
Description: The Lubben Social Network Scale (LSNS) was designed to measure perceived social support received from family and friends. The LSNS-Revised includes 12 items with scores ranging from 0-60 with higher scores indicating greater perceived social support.
Time Frame: One year
Reporting Status: Not Posted

13. Secondary Outcome: Level of Hospital Mobility
Description: All patients will wear a StepWatch throughout the hospitalization to document the level of mobility attained by each patient. The StepWatch is a ankle worn pedometer that documents number of steps taken and when they were taken.
Time Frame: Average one week
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Intensive | Friendly Visit
All-Cause Mortality (participants affected / at risk) | 10/60 | 9/68
Serious Adverse Events (participants affected / at risk) | 36/60 | 27/68
Other Adverse Events (participants affected / at risk) | 11/60 | 24/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intensive (N=60) | Friendly Visit (N=68)
Emergency Department visits (General disorders) | 36 (37) | 27 (41) — Visit to ED after initial hospital stay over a 6 month period
Rehospitalization (General disorders) | 36 (38) | 27 (36) — Readmission to the hospital in the 6-month period after the initial hospitalization
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intensive (N=60) | Friendly Visit (N=68)
skin irritation (General disorders) | 11 | 24 — Skin irritation at site for step watch

LIMITATIONS AND CAVEATS:
Study recruitment did not meet the calculated sample size target of 258 participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-02-05): https://cdn.clinicaltrials.gov/large-docs/03/NCT02674503/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-25): https://cdn.clinicaltrials.gov/large-docs/03/NCT02674503/SAP_001.pdf
  • Informed Consent Form (2017-10-25): https://cdn.clinicaltrials.gov/large-docs/03/NCT02674503/ICF_002.pdf